CLINICAL TRIAL: NCT01936675
Title: Myocardial Infarction Genes (MI-GENES) Study - Using Genomic Data to Refine Risk Assessment for Heart Attack
Brief Title: Myocardial Infarction Genes (MI-GENES) Study
Acronym: MI-GENES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Principal Investigator, Iftikhar J. Kullo, Professor of Medicine, Division of Cardiovascular Diseases, Department of Internal Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-001727; U01HG006379 (NIH)
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Coronary Artery Disease; Myocardial Infarction; Genomic Risk Communication
Keywords: Coronary Artery Disease; Myocardial Infarction; Genomic Risk Communication; Risk Stratification
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Framingham Risk Score (No Intervention): Patients in this arm will receive their Framingham Risk Score of having a heart attack.
- Framingham and Genetic Risk Score (Active Comparator): Patients in this arm will receive their Framingham Risk Score as well as their Genetic Risk Score of having a heart attack.
  Interventions: Other: Genetic Risk Score

INTERVENTIONS:
Other: Genetic Risk Score — Patients in this arm will receive their genetic-informed risk for having a heart attack.
  Arms: Framingham and Genetic Risk Score

SUMMARY:
This study is being done to better understand how genetic information might improve assessment of heart attack risk.

DETAILED DESCRIPTION:
This study aims to randomize patients to 2 arms. The first arm will receive the conventional Framingham risk score for coronary heart disease while the intervention arm will receive the genetics-informed risk for coronary artery disease.

The investigators will assess baseline blood lipid levels and follow the 2 arms up to 6 months after randomization. Primary endpoint is change in LDL levels between the 2 arms. Secondary outcomes include blood pressure control, weight, smoking cessation, and other lifestyle modifications.

This trial will help us understand whether coronary artery disease risk derived from genetic information would have a significant impact on patients' perception of coronary artery disease risk and motivate healthy lifestyle modifications that reduce their long term risk.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 45-70 years
* Patients who have participated in the Mayo Clinic Biobank or a previous research study at Mayo Clinic
* Patients who live in Southeast Minnesota

Exclusion Criteria:

* Taking statin or other lipid lowering medications
* Patients with a history of myocardial infarction, coronary artery disease, or other atherosclerotic medical conditions

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in serum LDL-cholesterol level | at 6 months post disclosure of CAD risk

SECONDARY OUTCOMES:
Change in HDL-cholesterol | at 6 months post disclosure of CAD risk
Change in systolic blood pressure measurements | at 6 months post disclosure of CAD risk
Change in fasting blood glucose measurements | at 6 months post disclosure of CAD risk
Number of Subjects Who Initiated Treatment with Statin Medications | at 6 months post disclosure of CAD risk
Number of Subjects Who Used the Patient Portal at One Year | at 6 months post disclosure of CAD risk
Shared decision making (as assessed by survey) | Immediately after risk disclosure
Physician visit satisfaction (as assessed by survey) | Immediately after risk disclosure
Genetic counseling satisfaction and perceived personal control (as assessed by survey) | Immediately after risk disclosure
Body mass index measurements | at 6 months post disclosure of CAD risk
Waist circumference | at 6 months post disclosure of CAD risk
Blood pressure | at 6 months post disclosure of CAD risk
Dietary fat intake (assessed by survey) | at 6 months post disclosure of CAD risk
Physical activity (assessed by survey) | at 6 months post disclosure of CAD risk
Smoking cessation | at 6 months post disclosure of CAD risk
Anxiety (assessed by survey) | at 6 months post disclosure of CAD risk
Rating of test results information (assessed by survey) | Immediately after risk disclosure and 6 months afterwards
Understanding of genetic risk or family history risk (assessed by survey) | Immediately after risk disclosure and 6 months afterwards
Reaction to test results information (assessed by survey) | Immediately after risk disclosure
Perceived risk (assessed by survey) | Immediately after risk disclosure and 6 months afterwards
Intention to change (assessed by survey) | 3 months after risk disclosure
Recall and measure of locus control (assessed by survey) | 3 months after risk disclosure
Motivation and perceptions (assessed by survey) | 3 months after risk disclosure
Attitudes towards genome sequencing (assessed by survey) | 3 and 6 months after risk disclosure
Impact of events scale (assessed by survey) | 3 and 6 months after risk disclosure
Genetic knowledge (assessed by survey) | at enrollment and 6 months after risk disclosure
Attitude toward genetic testing (assessed by survey) | 6 months after risk disclosure
Decisional regret and treatment beliefs (assessed by survey) | 6 months after risk disclosure
Use of internet, electronic health record, social networks, and information sharing (assessed by survey) | 3 and 6 months after risk disclosure

CONTACTS AND LOCATIONS:
Overall Officials: Iftikhar Kullo, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ding K, Bailey KR, Kullo IJ. Genotype-informed estimation of risk of coronary heart disease based on genome-wide association data linked to the electronic medical record. BMC Cardiovasc Disord. 2011 Nov 3;11:66. doi: 10.1186/1471-2261-11-66. PMID 22151179
- [Result] Robinson CL, Jouni H, Kruisselbrink TM, Austin EE, Christensen KD, Green RC, Kullo IJ. Disclosing genetic risk for coronary heart disease: effects on perceived personal control and genetic counseling satisfaction. Clin Genet. 2016 Feb;89(2):251-7. doi: 10.1111/cge.12577. Epub 2015 Mar 23. PMID 25708169
- [Result] Kullo IJ, Jouni H, Olson JE, Montori VM, Bailey KR. Design of a randomized controlled trial of disclosing genomic risk of coronary heart disease: the Myocardial Infarction Genes (MI-GENES) study. BMC Med Genomics. 2015 Aug 15;8:51. doi: 10.1186/s12920-015-0122-0. PMID 26271327
- [Result] Kullo IJ, Jouni H, Austin EE, Brown SA, Kruisselbrink TM, Isseh IN, Haddad RA, Marroush TS, Shameer K, Olson JE, Broeckel U, Green RC, Schaid DJ, Montori VM, Bailey KR. Incorporating a Genetic Risk Score Into Coronary Heart Disease Risk Estimates: Effect on Low-Density Lipoprotein Cholesterol Levels (the MI-GENES Clinical Trial). Circulation. 2016 Mar 22;133(12):1181-8. doi: 10.1161/CIRCULATIONAHA.115.020109. Epub 2016 Feb 25. PMID 26915630
- [Derived] Naderian M, Hamed ME, Vaseem AA, Norland K, Dikilitas O, Teymourzadeh A, Bailey KR, Kullo IJ. Effect of Disclosing a Polygenic Risk Score for Coronary Heart Disease on Adverse Cardiovascular Events. Circ Genom Precis Med. 2025 Apr;18(2):e004968. doi: 10.1161/CIRCGEN.124.004968. Epub 2025 Mar 28. PMID 40151934
- [Derived] Brown SN, Jouni H, Kullo IJ. Electronic health record access by patients as an indicator of information seeking and sharing for cardiovascular health promotion in social networks: Secondary analysis of a randomized clinical trial. Prev Med Rep. 2019 Jan 14;13:306-313. doi: 10.1016/j.pmedr.2018.12.011. eCollection 2019 Mar. PMID 30792945
- [Derived] Brown SN, Jouni H, Marroush TS, Kullo IJ. Effect of Disclosing Genetic Risk for Coronary Heart Disease on Information Seeking and Sharing: The MI-GENES Study (Myocardial Infarction Genes). Circ Cardiovasc Genet. 2017 Aug;10(4):e001613. doi: 10.1161/CIRCGENETICS.116.001613. PMID 28779015
- [Derived] Jouni H, Haddad RA, Marroush TS, Brown SA, Kruisselbrink TM, Austin EE, Shameer K, Behnken EM, Chaudhry R, Montori VM, Kullo IJ. Shared decision-making following disclosure of coronary heart disease genetic risk: results from a randomized clinical trial. J Investig Med. 2017 Mar;65(3):681-688. doi: 10.1136/jim-2016-000318. Epub 2016 Dec 19. PMID 27993947